CLINICAL TRIAL: NCT04402827
Title: Differences in Susceptibility to SARS CoV-2 Infection According to ACE2 and CD26 Receptors, Specific CD4/CD8 T Cell Response to Viral Peptides, and KIR Receptors Among Health Care Workers Highly Exposed to Patients With COVID-19 Diagnosis.
Brief Title: Different Susceptibility to SARS CoV-2 Infection Among Health Care Workers Highly Exposed to COVID-19.
Acronym: CoVEX
Status: Completed | Type: Observational
Sponsor: Asociacion para el Estudio de las Enfermedades Infecciosas (Network)
Responsible Party: Sponsor
Other Study IDs: EC 162/20
Record Dates: First submitted 2020-05-23; First posted 2020-05-27 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Health Care Worker Patient Transmission; Receptor Site Alteration; Susceptibility, Disease; Immune Response
Keywords: coronavirus, susceptibility, transmission, HCW
MeSH Terms: conditions — Disease Susceptibility; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: HCW highly exposed (defined as more than 15 days of continued personal attention in ICU, anaesthesia, or Infectious Diseases wards) to patients with a diagnosis of COVID-19 (PCR confirmed), who remained asymptomatic and with a negative serology (IgM and IgG negative). Transient entry or stay in the zone (kitchen personnel, rehab members,...) will be not included.
  Interventions: Diagnostic Test: Susceptibility to infection
- Controls: HCW highly exposed to PCR-confirmed patients with a diagnosis of COVID-19, as defined above, matched by age and sex, who had suffered confirmed SARS CoV-2 disease (positive PCR or after, positive IgG)
  Interventions: Diagnostic Test: Susceptibility to infection

INTERVENTIONS:
Diagnostic Test: Susceptibility to infection — ACE2 and CD26 receptor study: After genomic DNA extraction and quantification using a NanoDrop-1000, 14 ACE2 SNPs (rs1978124, rs2048683, rs2074192, rs2106809, rs2285666, rs233575, rs4240157, rs4646142, rs4646155, rs4646156, rs4646188, rs4830542, rs6632677, and rs879922) will be studied. In addition, one CD26 (DPP4) SNP (rs7608798) will be analysed (qualitative measure).
  SARS-CoV-2 CD4/CD8 T cell response: SARS-CoV-2 peptides (Prot-S, Pros-N and Port-M) will be used to activate CD4 and CD8 T cells. Cytokines released, such as IFNg, TNFa, IL4, IL17A, and IL2, from each cell subset will be measured by flow cytometry (quantitative measure).
  KIR characterization: Characterization of the presence of 14 genes plus 2 pseudogenes of KIR gene family (qualitative genotyping) by PCR, mRNA expression profiling (quantitative measures) by RT-PCR, and phenotyping of human NK cells analyzing different KIR receptors (quantitative measure) by flow cytometry, will be analyzed.
  Other Names: KIR measurements

SUMMARY:
The primary objective of this study is to establish differences in susceptibility to SARS CoV-2 infection among health care workers (HCW) highly exposed to patients with COVID-19 diagnosis. To ascertain this issue, we evaluated:

* Changes in receptor polymorphism (ACE2 and CD26 receptor study.
* SARS-CoV-2 CD4/CD8 T cell response (CTL)
* Different KIR phenotypes

DETAILED DESCRIPTION:
Only 24% of health care workers (HCW) had developed inmunological response to SARS CoV-2 infection in one centre attending thousands of COVID-19 patients, and with shorteness of personal protective equipments. Our hypothesis is that this relatively low number of infected HCW could be secondary to:

1. Differences in susceptibility to infection mediated by changes in viral receptors. Thus, it is important to characterize and genotyping the main receptor for SARS-CoV-2, ACE2, and other related receptor, such as CD26.
2. Increased cellular immune response, offering cross-immunity against SARS CoV-2 infection by previous exposure to other coronavirus or respiratory pathogens. A specific CD4/CD8 T cell response to viral peptides could respond this question
3. Specific KIR phenotypes (Killer Immunoglobulin-like Receptors): Natural killer cells (NK) response to alterations of class I HLA molecules presented in infected cells. An increase in class I HLA expression could lead to an increase in NK activation by increasing its ability to produce IFN-gamma.

ELIGIBILITY:
Inclusion criteria

* HCW older than 18 years
* Highly exposed to COVID-19 according to the definition
* Negative (cases) or positive (controls) serology against SARS-CoV-2 infection Exclusion criteria
* Presence of any disease / treatment which could alter the susceptibility (corticoid therapy, chemotherapy, monoclonal antibodies)
* Pregnancy

High exposure definition: direct and continued care of COVID-19 diagnosed patients for 2 weeks or more, without aerosol- generating procedures, with inappropriate personal protective equipment (PPE), or unprotected exposure to patients with COVID-19 during aerosol-generating procedures.

The definition of appropriate PPE was based on previous recommendations. The absence of any part of the PPE constituted an unprotected exposure. We defined the following as aerosol-generating procedures: airway suction, application of a high-flow O2 instrument, bronchoscopy, endotracheal intubation, tracheostomy, nebulizer treatment, sputum induction, positive pressure ventilation, manual ventilation and cardiopulmonary resuscitation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Cases: HCW highly exposed to COVID-19 diagnosed patients (see definition) who remained free of symptoms of disease and had a negative serology against SARS-CoV-2 (both IgG and IgM)
  * Controls: HCW highly exposed to COVID-19 diagnosed patients who had suffered the infection and/or had presence of antibodies in the serological test, paired by sex and age (5 year interval)
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Susceptibility to SARS CoV-2 infection according to ACE2 receptor | 1 month
  ACE2 analysis
Cellular immune response to SARS CoV-2 infection | 1 month
  Activation of CD4-CD8 by viral peptides
Susceptibility to infections according to KIR phenoytpes | 2 months
  Analysis of KIR in NK cells

SECONDARY OUTCOMES:
Characteristics of exposure in time and intensity of HCW with SARS CoV-2 infection | 1 month
  Survey
Cellular immune response in HCW with positive IgG against SARS CoV-2 | 1 month
  Activation of CD4-CD8 by viral peptides

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Casado, MD, PhD, Principal Investigator — Ramon y Cajal Physician
Locations (1):
- Hospital Ramon y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Data about receptors could be shared with other investigators about the susceptiblity to SARS CoV-2 However, KIR phenotypes should be shared after ethical comitee approval

REFERENCES:
- [Derived] Vizcarra P, Haemmerle J, Velasco H, Velasco T, Fernandez-Escribano M, Vallejo A, Casado JL. BNT162b2 mRNA COVID-19 vaccine Reactogenicity: The key role of immunity. Vaccine. 2021 Dec 17;39(51):7367-7374. doi: 10.1016/j.vaccine.2021.10.074. Epub 2021 Nov 11. PMID 34802792